CLINICAL TRIAL: NCT07165249
Title: Positional Release Technique Versus Muscle Energy Technique For Patients With Non-Specific Low Back Pain With Facet Joint Restriction
Brief Title: PRT vs MET in Non-Specific Low Back Pain With Facet Restriction
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palestine Ahliya University (Other)
Responsible Party: Principal Investigator, Azzam Alarab, Assistant Professor Chairperson, Department of Medical Sciences - Master's, Palestine Ahliya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PalestineAhliyaU
Record Dates: First submitted 2025-08-25; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Non Specific Low Back Pain; Muscle Energy Technique
Keywords: Muscle energy; PRT; Non specific low back pain

STUDY DESIGN:
Intervention Model Description: Group A (PRT): Positional Release Technique - 3 sessions/week for 4 weeks with hot pack co-intervention Group B (MET): Muscle Energy Technique - 3 sessions/week for 4 weeks with hot pack co-intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm 1- Group A (PRT): Positional Release Technique (Experimental): 3 sessions/week for 4 weeks with hot pack co-intervention.
  Interventions: Behavioral: Positional release technique (PRT)
- arm2- Group B (MET): Muscle Energy Technique (Experimental): 3 sessions/week for 4 weeks with hot pack co-intervention.
  Interventions: Behavioral: Muscle energy technique

INTERVENTIONS:
Behavioral: Positional release technique (PRT) — Group A (PRT): Patients lay prone for the application of the hot pack. PRT was then applied to the erector spinae muscles. The therapist identified tender points and passively positioned the patient into a position of comfort, typically involving lateral trunk flexion toward the symptomatic side. Each session involved three 90-second holds per tender point. PRT procedures followed standardized positioning principles as described in previous literature.
  Arms: arm 1- Group A (PRT): Positional Release Technique
Behavioral: Muscle energy technique — Group B (MET): Following the hot pack application, patients were assessed for segmental dysfunction via palpation of lumbar transverse processes in prone position. MET was applied using isometric contractions aimed at correcting lumbar rotational or side-bending dysfunctions. Each contraction was held for 7-10 seconds, followed by a passive stretch. The technique was repeated for 3-5 cycles per session.
  Arms: arm2- Group B (MET): Muscle Energy Technique

SUMMARY:
Objective:The study aimed to compare the effectiveness of Positional Release Technique (PRT) and Muscle Energy Technique (MET) in reducing pain and improving outcomes for patients suffering from non-specific low back pain (NSLBP).

Materials and Methods: Thirty-six patients between the ages of 25 and 50, all referred by an orthopedic surgeon for treatment of non-specific low back pain (NSLBP), were enrolled in the study. Participants were randomly allocated into two groups (n=18 per group) using a computer-generated randomization sequence. However, details regarding allocation concealment and blinding of participants or assessors were not specified, which may influence the risk of bias. Group A received Positional Release Technique (PRT), while Group B received Muscle Energy Technique (MET). Prior to each treatment session, both groups received a standardized 15-minute hot pack application as a co-intervention to promote muscle relaxation and ensure consistency across interventions. Pain intensity was assessed using the Visual Analogue Scale (VAS), and functional outcomes were measured with the Roland-Morris Disability Questionnaire (RMQ). Participants in both groups attended three physiotherapy sessions per week over a four-week treatment period.

DETAILED DESCRIPTION:
1. Study Identification

   Official Title:

   Positional Release Technique Versus Muscle Energy Technique for Patients with Non-Specific Low Back Pain With Facet Joint Restriction

   Brief Title:

   PRT vs MET in Non-Specific Low Back Pain

   Study Type:

   Interventional (Clinical Trial)

   Phase:

   Not Applicable
2. Study Description

   Brief Summary:

   This study aimed to compare the effectiveness of Positional Release Technique (PRT) and Muscle Energy Technique (MET) in reducing pain and improving outcomes for patients suffering from non-specific low back pain with suspected facet joint dysfunction. Thirty-six patients were randomized into two groups and received treatment for 4 weeks, 3 sessions per week. Pain intensity (VAS) and functional disability (Roland-Morris Questionnaire) were assessed pre- and post-intervention.
3. Study Design

   Allocation: Randomized

   Intervention Model: Parallel Assignment

   Masking: None (Open Label)

   Primary Purpose: Treatment
4. Conditions & Interventions

   Condition:

   Non-Specific Low Back Pain (NSLBP)

   Interventions:

   Group A (PRT): Positional Release Technique - 3 sessions/week for 4 weeks with hot pack co-intervention.

   Group B (MET): Muscle Energy Technique - 3 sessions/week for 4 weeks with hot pack co-intervention.
5. Outcome Measures

   Primary Outcome Measures:

   Pain intensity (VAS) - Baseline and after 4 weeks.

   Functional disability (Roland-Morris Questionnaire, RMQ) - Baseline and after 4 weeks.
6. Eligibility

   Ages Eligible for Study: 25-50 years

   Sexes Eligible for Study: All

   Inclusion Criteria: Chronic NSLBP >3 months, suspected facet joint dysfunction.

   Exclusion Criteria: History of spinal surgery, vertebral fracture, osteoporosis, inflammatory/metabolic bone disease, spondylolisthesis.
7. Enrollment

   Enrollment: 36 participants (actual)
8. Locations

Maqassed Hospital, East Jerusalem, Palestine

ELIGIBILITY:
Inclusion criteria:

* Participants in the age category of 25 to 50 years old.
* both male and female, with a diagnosis of low back pain (LBP), with or without referred leg pain.
* chronic LBP lasting more than three months.

Exclusion criteria:

* Osteoporosis.
* bone disease.
* Spondylolisthesis.
* History of vertebral fracture.
* History of spinal surgery.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-02 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
VAS - Baseline and after 4 weeks. Functional disability (Roland-Morris Questionnaire, RMQ) - Baseline and after 4 weeks. | 4 weeks
  A popular instrument for measuring pain is the visual analogue scale (VAS). Typically, it's a 10-cm line with the words "worst pain imaginable" at one end and "no pain" at the other. In order to quantify their level of pain, patients mark the line, and the distance from "no pain" serves as a proxy for pain
RMQ | 4 weeks
  It asks about 24 different activities and functions that could be impacted by back pain. Patients indicate if they now find it difficult to be active owing to back discomfort by answering "yes" or "no" to each topic. The total number of "yes" responses is added up to determine the score; a higher score denotes a larger disability

CONTACTS AND LOCATIONS:
Locations (1):
- Palestine Ahliya University, Bethlehem, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared with other researchers, as there are no plans for data sharing.